CLINICAL TRIAL: NCT01274338
Title: A Phase III Randomized Study of Adjuvant Ipilimumab Anti-CTLA4 Therapy Versus High-Dose Interferon a-2b for Resected High-Risk Melanoma
Brief Title: Ipilimumab or High-Dose Interferon Alfa-2b in Treating Patients With High-Risk Stage III-IV Melanoma That Has Been Removed by Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02649; NCI-2011-02649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000692568; ECOG-E1609; E1609; E1609 (Other: ECOG-ACRIN Cancer Research Group); E1609 (Other: CTEP); P50CA121973 (NIH); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2011-01-08; First posted 2011-01-11 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Melanoma of Unknown Primary; Recurrent Melanoma; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm A (age >= 18, high-dose ipilimumab) (Experimental): Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity. (closed accrual as of 4/4/14) (adult accrual has completed to Arms A, B, and C as of 8/15/2014)
  Interventions: Biological: Ipilimumab; Other: Quality-of-Life Assessment
- Arm B (age >= 18, recombinant interferon alfa-2b) (Experimental): Patients receive high-dose recombinant interferon alpha-2b IV on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alpha-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity. (adult accrual has completed to Arms A, B, and C as of 8/15/2014)
  Interventions: Other: Quality-of-Life Assessment; Biological: Recombinant Interferon Alfa-2b
- Arm C (age >= 18, low-dose ipilimumab) (Experimental): Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cyclees in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity. (adult accrual has completed to Arms A, B, and C as of 8/15/2014)
  Interventions: Biological: Ipilimumab; Other: Quality-of-Life Assessment
- Arm D (age 12-17, high-dose ipilimumab) (Experimental): Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab
- Arm E (ages 12-17, recombinant interferon alfa-2b) (Experimental): Patients receive high-dose recombinant interferon alpha-2b IV on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alpha-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity. (ages 12-17)
  Interventions: Biological: Recombinant Interferon Alfa-2b
- Arm F (ages 12-17, low-dose ipilimumab) (Experimental): Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity. (ages 12-17)
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm A (age >= 18, high-dose ipilimumab); Arm C (age >= 18, low-dose ipilimumab); Arm D (age 12-17, high-dose ipilimumab); Arm F (ages 12-17, low-dose ipilimumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm A (age >= 18, high-dose ipilimumab); Arm B (age >= 18, recombinant interferon alfa-2b); Arm C (age >= 18, low-dose ipilimumab)
Biological: Recombinant Interferon Alfa-2b — Given IV and SC
  Other Names: Alfatronol; Bioferon; Bioferon (TM); Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Arm B (age >= 18, recombinant interferon alfa-2b); Arm E (ages 12-17, recombinant interferon alfa-2b)

SUMMARY:
This randomized phase III trial studies ipilimumab to see how well it works compared to high-dose interferon alfa-2b in treating patients with high-risk stage III-IV melanoma that has been removed by surgery. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Interferon alfa-2b may interfere with the growth of tumor cells and slow the growth of melanoma and other cancers. It is not yet known whether ipilimumab is more effective than interferon alfa-2b in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate recurrence-free survival (RFS) between patients randomized to receive post-operative adjuvant ipilimumab given at either 10 mg/kg (high dose ipilimumab; HIP) or 3 mg/kg (low dose ipilimumab: LIP) versus those randomized to receive high-dose interferon alfa-2b (HDI) utilizing a hierarchical design assessing HIP versus HDI first and LIP versus HDI second (if the first comparison is significant).

II. To evaluate overall survival (OS) between patients randomized to receive post-operative adjuvant ipilimumab given at either 10 mg/kg (HIP) or 3 mg/kg (LIP) versus those randomized to receive HDI utilizing a hierarchical design assessing HIP versus HDI first and LIP versus HDI second (if the first comparison is significant).

SECONDARY OBJECTIVES:

I. To evaluate safety and tolerability of post-operative adjuvant ipilimumab therapy given at either 10 mg/kg (HIP) or 3 mg/kg (LIP).

II. Among patients enrolled by Clinical Community Oncology programs (CCOPs), to compare the global quality of life (QOL) between the ipilimumab arms versus HDI using Functional Assessment of Cancer Therapy (FACT)-General (G) form and to evaluate the effect of treatment-related side effects that may have an impact on the health-related domains of QOL using Functional Assessment of Chronic Illness Therapy (FACIT)-diarrhea (D) and FACT-biological response modifiers (BRM).

OUTLINE: Patients age >= 18 are randomized to Arms A, B, or C and patients ages 12-17 are randomized to Arms D, E, or F.

ARM A: Patients receive induction high-dose ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity. (closed accrual as of 4/4/14) (adult accrual has completed to Arms A, B, and C as of 8/15/2014)

ARM B: Patients receive induction high-dose recombinant interferon alfa-2b IV over 20 minutes on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alfa-2b subcutaneously (SC) on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity. (adult accrual has completed to Arms A, B, and C as of 8/15/2014)

ARM C: Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity. (adult accrual has completed to Arms A, B, and C as of 8/15/2014)

ARM D: Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive induction high-dose recombinant interferon alfa-2b IV over 20 minutes on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alfa-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity

ARM F: Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 90 days for a maximum of 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have disease-free status documented by a complete physical examination and imaging studies within 4 weeks prior to randomization; imaging studies must include a total body positron emission tomography (PET)-computed tomography (CT) scan (with or without brain) and brain magnetic resonance imaging (MRI) or CT (if MRI is contraindicated); if PET-CT cannot be done, CT of neck, chest, abdomen, and pelvis should be done

  * If for some reason a CT cannot be done, an MRI may be done instead; any other imaging studies if performed (eg, bone scan) must show no evidence of disease
* Patients must have primary cutaneous melanoma that belong to one of the following American Joint Commission on Cancer (AJCC) stages (2009 AJCC Melanoma Staging System):

  * Stage IIIB

    * T1-4b N1a M0
    * T1-4b N2a M0
    * T1-4b N1b M0
    * T1-4b N2b M0
    * T1-4b N2c M0
  * Stage IIIC

    * T1-4b N1b M0
    * T1-4b N2b M0
    * T1-4b N2c M0
    * Any T N3 M0
  * Stage IV

    * M1a
    * M1b
    * NOTE: patients with stage IV melanoma must have normal lactate dehydrogenase (LDH) and either distant skin, subcutaneous, lymph node, or lung metastases, but no other visceral metastases in order to be eligible; for patients with resected stage IV melanoma, LDH within the institutional upper limit of normal (ULN) must be documented within 4 weeks prior to randomization
* Patients with disease recurrence after adequate surgical excision of the original primary cutaneous/unknown primary melanoma are allowed even if they don't fit the strict staging criteria, but only as follows:

  * Recurrence in a regional lymph node basin after a prior complete lymph node dissection; relapsed disease must be completely surgically resected with free margins
  * Recurrence in the form of in-transit or satellite metastases or distant skin/subcutaneous, nodal, or lung metastases that are completely surgically resected with free margins
  * Recurrence in a regional lymph node basin; relapsed disease must be completely surgically resected with free margins
* Patients with unknown primary melanoma (Tx) who present with cutaneous, subcutaneous, nodal and/or lung metastases that are completely surgically resected with free margins are allowed; these patients are allowed even if they don't fit the strict staging criteria; for stage IV patients LDH within the institutional ULN must be documented within 4 weeks prior to randomization (M1c is not eligible)

  * NOTE: all subjects should be classified as IIIB, IIIC, M1a or M1b including subjects with disease recurrence after adequate surgical excision of the original primary melanoma; that is the treating team/physician investigator should review an overall TNM status (that includes primary tumor presentation and disease recurrence status) and provide a designation of IIIB, IIIC, M1a or M1b
* Patients must be randomized within 84 days (12 weeks) of surgical resection; if more than one surgical procedure is required to render the patient disease-free, the patient must be randomized within 12 weeks of the last surgery

  * NOTE: patients with clinically positive lymph nodes for melanoma involvement or those with positive lymph nodes identified through lymphoscintigraphic and/or dye lymphographic techniques in the groin, axilla, or neck should have additional lymphadenectomy in those sites; the complete lymph node dissection procedure would be considered as the last surgery in counting the 84 days unless a subsequent surgical procedure(s) was clinically required to ensure the disease free status
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Given that serious adverse events may occur with ipilimumab and IFN-alpha and that these may impact a patient's wellbeing, it is possible that the occurrence of other serious adverse events (SAEs) may seriously impact an underlying state of mental depression and lead to suicidal ideation; therefore, patients should be carefully screened for depression at baseline and if there are indications or a history of depression it is strongly recommended that these patients be closely followed together with behavioral health or psychiatric medical support; patients with an established diagnosis of depression that, in the assessment of the investigator may make the administration of IFN-alpha or ipilimumab hazardous, should not be enrolled on this protocol; the risks and benefits of being treated with standard adjuvant IFN-alpha should be weighed very carefully in consultation with behavioral health or psychiatry
* Due to the possible effect of treatment with ipilimumab on the immunologic response to infectious disease vaccines, patients must not have had any infectious disease vaccination (e.g., standard influenza, H1N1 influenza, pneumococcal, meningococcal, tetanus toxoid) within 4 weeks prior to randomization
* WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of ipilimumab or HDI, in such a manner that the risk of pregnancy is minimized; women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential

  * Men of fathering potential and WOCBP must be using an adequate method of contraception to avoid conception/pregnancy throughout the study and for up to 26 weeks after the last dose of ipilimumab or HDI in such a manner that the risk of pregnancy is minimized; men or WOCBP who are unwilling or unable to strictly follow this requirement are not eligible
  * WOCBP are not eligible if they satisfy any of the following:

    * A positive pregnancy test at baseline
    * Pregnant or breastfeeding
* White blood cell (WBC) >= 3,000/uL (obtained within 4 weeks prior to randomization)
* Absolute neutrophil count (ANC) >= 1,500/uL (obtained within 4 weeks prior to randomization)
* Platelets >= 100 x 10^3/uL (obtained within 4 weeks prior to randomization)
* Hemoglobin >= 10 g/dL (obtained within 4 weeks prior to randomization)
* Serum creatinine =< 1.5 mg/dL (obtained within 4 weeks prior to randomization)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN (obtained within 4 weeks prior to randomization)
* Serum bilirubin =< 1.5 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL) (obtained within 4 weeks prior to randomization)
* No active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C due to the unknown effects of ipilimumab; patients must have negative testing for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) within 4 weeks prior to randomization

Exclusion Criteria:

* Patients must not have received any adjuvant treatment (chemotherapy, biotherapy, or limb perfusion) after the resection(s) that make(s) them eligible for this trial

  * NOTE: previous radiation therapy, including after the surgical resection, is allowed as long as 21 days have elapsed between the radiation and initiation of this adjuvant systemic therapy
* Prior treatment with anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) monoclonal antibodies or prior CTLA-4 inhibitor or agonist or prior clusters of differentiation (CD)137 agonist or prior interferon-alfa is not allowed; other forms of prior treatment for melanoma (e.g., aldesleukin [IL-2], anti-tumor vaccine, chemotherapy) are allowed if given before the resection(s) that make(s) the patient eligible for this trial, but these must have been completed at least 4 weeks prior to randomization
* Patients must not have an active infection requiring current treatment with parenteral antibiotics
* Patients must not have other significant medical, surgical, or psychiatric conditions or require any medication or treatment that in the opinion of the investigator may interfere with compliance, make the administration of ipilimumab or HDI hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea; patients with a baseline of frequent diarrhea (e.g. irritable bowel syndrome) are not eligible because of the difficulty in interpreting later expected GI toxicities that may lead to suboptimal management and complications
* Patients must not have a documented history of inflammatory bowel disease (including ulcerative colitis and Crohn's disease) or diverticulitis (history of diverticulosis is allowed)
* Patients must not have autoimmune disorders or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids; a history of occasional (but not continuous) use of steroid inhalers is allowed; replacement doses of steroids for patients with adrenal insufficiency are allowed; patients who discontinue use of these classes of medication for at least 2 weeks prior to randomization are eligible if, in the judgment of the treating physician investigator, the patient is not likely to require resumption of treatment with these classes of drugs during the study

  * Exclusion from this study also includes patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjogren's syndrome, autoimmune vasculitis [e.g., Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and Myasthenia Gravis); other central nervous system (CNS) autoimmune disease (e.g., poliomyelitis, multiple sclerosis)
  * Patients with autoimmune hypothyroid disease or type I diabetes on replacement treatment are eligible
* Patients must not be prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness; this is due to concerns about subject safety and compliance with study procedures
* Patients who have other current malignancies are not eligible; patients with other malignancies are eligible if they have been continuously disease free for > 5 years prior to the time of randomization; patients with prior history at any time of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or melanoma in situ are eligible; patients with prior history of basal or squamous skin cancer are eligible; patients who have had multiple primary melanomas are eligible
* Women must not be pregnant or breast-feeding due to the unknown effects of ipilimumab and HDI on conception and the fetus; all females of childbearing potential must have a blood test or urine study during screening to rule out pregnancy

  * NOTE: a woman of childbearing potential (WOCBP) is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); post-menopause is defined as:

    * Amenorrhea >= 12 consecutive months without another cause, or
    * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1673 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (939):
- United States (930):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin Cancer Care Inc, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - AdventHealth Daytona Beach, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Cancer Center of Putnam, Palatka, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Martin Medical Center, Stuart, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Martin Hospital South, Stuart, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - York Hospital, York Village, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Mission Hospital McDowell, Marion, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Health Sciences North, Greater Sudbury, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

REFERENCES:
- [Derived] McLouth LE, Zheng Y, Smith S, Hodi FS, Rao UN, Cohen GI, Amatruda TT, Dakhil SR, Curti BD, Nakhoul I, Chandana SR, Bane CL, Marinier DE, Lee SJ, Sondak VK, Kirkwood JM, Tarhini AA, Wagner LI. Patient-reported tolerability of adjuvant ipilimumab (3 or 10 mg/kg) versus high-dose interferon alfa-2b for resected high-risk stage III-IV melanoma in phase III trial E1609. Qual Life Res. 2023 Jan;32(1):183-196. doi: 10.1007/s11136-022-03226-8. Epub 2022 Aug 27. PMID 36029412
- [Derived] Saad M, Lee SJ, Tan AC, El Naqa IM, Hodi FS, Butterfield LH, LaFramboise WA, Storkus W, Karunamurthy AD, Conejo-Garcia J, Hwu P, Streicher H, Sondak VK, Kirkwood JM, Tarhini AA. Enhanced immune activation within the tumor microenvironment and circulation of female high-risk melanoma patients and improved survival with adjuvant CTLA4 blockade compared to males. J Transl Med. 2022 Jun 3;20(1):253. doi: 10.1186/s12967-022-03450-3. PMID 35659704
- [Derived] Johnson DB, Friedman DL, Berry E, Decker I, Ye F, Zhao S, Morgans AK, Puzanov I, Sosman JA, Lovly CM. Survivorship in Immune Therapy: Assessing Chronic Immune Toxicities, Health Outcomes, and Functional Status among Long-term Ipilimumab Survivors at a Single Referral Center. Cancer Immunol Res. 2015 May;3(5):464-9. doi: 10.1158/2326-6066.CIR-14-0217. Epub 2015 Feb 3. PMID 25649350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1673 patients, including 1670 adult patients and 3 pediatric patients, were accrued between May 25, 2011 and July 26, 2016. Accrual of adult patients were completed on August 15, 2014. The study was reactivated to accrue pediatric patients on September 23, 2014.
Groups:
- Arm A (HIP): Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (HDI): Patients receive high-dose recombinant interferon alpha-2b IV on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alpha-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity.
- Arm C (LIP): Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm D (HIP; Pediatric): Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity. (ages 12-17)
- Arm E (HDI; Pediatric): Patients receive high-dose recombinant interferon alpha-2b IV on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alpha-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity. (ages 12-17)
- Arm F (LIP; Pediatric): Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity. (ages 12-17)
Period: Overall Study
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP) | Arm D (HIP; Pediatric) | Arm E (HDI; Pediatric) | Arm F (LIP; Pediatric)
Started | 511 | 636 | 523 | 1 | 1 | 1
Received Treatment | 503 | 520 | 516 | 1 | 1 | 1
Data Available for the FACT-G and FACT-BRM Analyses | 110 | 114 | 97 | 0 | 0 | 0
Data Available for FACIT-D Analysis | 109 | 114 | 97 | 0 | 0 | 0
Completed | 108 | 182 | 198 | 0 | 0 | 1
Not Completed | 403 | 454 | 325 | 1 | 1 | 0
Not completed — Lack of Efficacy | 72 | 108 | 116 | 0 | 0 | 0
Not completed — Adverse Event | 272 | 105 | 180 | 1 | 0 | 0
Not completed — Death | 8 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 99 | 17 | 0 | 0 | 0
Not completed — Did not start treatment | 8 | 116 | 7 | 0 | 0 | 0
Not completed — Alternative therapy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other complicating diseases | 0 | 3 | 1 | 0 | 0 | 0
Not completed — Treatment arm was suspended due to toxicity | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reason not reported | 12 | 21 | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP) | Arm D (HIP; Pediatric) | Arm E (HDI; Pediatric) | Arm F (LIP; Pediatric) | Total
Number analyzed (Participants) | 511 | 636 | 523 | 1 | 1 | 1 | 1673
Age, Continuous [Median (Full Range); unit: years] | 54 [18 to 60] | 54 [18 to 83] | 54 [19 to 80] | 15 [15 to 15] | 17 [17 to 17] | 17 [17 to 17] | 54 [15 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 241 | 195 | 1 | 1 | 0 | 607
  Male | 342 | 395 | 328 | 0 | 0 | 1 | 1066
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 20 | 16 | 0 | 0 | 0 | 44
  Not Hispanic or Latino | 484 | 591 | 488 | 1 | 1 | 1 | 1566
  Unknown or Not Reported | 19 | 25 | 19 | 0 | 0 | 0 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 3 | 0 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 0 | 0 | 0 | 5
  White | 497 | 620 | 510 | 1 | 1 | 1 | 1630
  More than one race | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 7 | 9 | 8 | 0 | 0 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS; Arm B [HDI] vs. Arm C [LIP])
Description: Recurrence-free survival is defined as the time from randomization to recurrence or death, whichever occurs first. The following criteria constitute the only acceptable evidence of disease recurrence.
  Lung and liver: Positive cytology or biopsy in the presence of a single new lesion or the appearance of multiple lesions consistent with metastatic disease.
  Central Nervous System: A positive brain CT or MRI scan or CSF cytology. Cutaneous, Subcutaneous and Lymph Node Recurrence: Positive cytology or biopsy in the presence of a single new lesion or the appearance of multiple lesions consistent with metastatic disease.
  Bone and Other Organs: Positive cytology or biopsy in the presence of a single new lesion or the appearance of multiple lesions consistent with metastatic disease identified on two different radiologic studies: i.e., positive nuclear bone scan or PET scan and contrast GI series or ultrasound, X-ray or CT of abdomen for abdominal disease.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for years 3-5 and then annually up to 8 years
Population: Concurrently randomized patients on Arms B and C
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm B (HDI) | Arm C (LIP)
Number analyzed (Participants) | 528 | 523
years | 2.5 [1.7 to 3.3] | 4.5 [2.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Arm B (HDI) vs Arm C (LIP); This study has a two-step hierarchical approach. In the first step, the low-dose Ipi (LIP) will be compared with HDI. If the low-dose Ipi is significantly better than HDI, then the high-dose Ipi will be compared with HDI as a second step. When comparing the two investigational treatment groups, the primary comparison will be an intent to treat analysis of recurrence free survival (RFS; First Co-primary Endpoint) and overall survival (OS; Second Co-primary Endpoint); Test type: Superiority; p = 0.065, Log Rank — This design provides at least 80% power at a one sided type I error rate of 0.003; Stratified logrank test

2. Primary Outcome: 5-year Overall Survival (OS) Rate (Arm B [HDI] vs. Arm C [LIP])
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for years 3-5
Population: Concurrently randomized patients on Arms B and C
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm B (HDI) | Arm C (LIP)
Number analyzed (Participants) | 528 | 523
proportion of participants | 0.67 [0.62 to 0.72] | 0.72 [0.68 to 0.76]
Statistical Analysis 1: Comparison: Arm B (HDI) vs Arm C (LIP); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This design will provide 80% power to detect the difference between the two arms at a one-sided type I error rate of 0.022; p = 0.044, Log Rank; Stratified logrank test

3. Primary Outcome: Recurrence-free Survival (RFS; Arm A [HIP] vs. Arm B [HDI])
Description: as for outcome 1
Time Frame: Assessed every 3 months for 2 years, then every 6 months for years 3-5 and then annually up to 8 years
Population: Concurrently randomized patients on Arms A and B
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A (HIP) | Arm B (HDI)
Number analyzed (Participants) | 511 | 478
years | 3.9 [2.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 2.4 [1.6 to 3.0]

4. Primary Outcome: 5-year Overall Survival (OS) Rate (Arm A [HIP] vs. Arm B [HDI])
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for years 3-5
Population: Concurrently randomized patients on Arms A and B
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (HIP) | Arm B (HDI)
Number analyzed (Participants) | 511 | 478
proportion of participants | 0.70 [0.65 to 0.74] | 0.65 [0.60 to 0.70]
Statistical Analysis 1: Comparison: Arm A (HIP) vs Arm B (HDI); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.289, Log Rank — If low dose Ipi (LIP) vs. HDI is significant for OS at the 2.2% level, then we will compare high dose Ipi (HIP) vs. HDI at the 2.2% level; Stratified logrank test

5. Secondary Outcome: Change in FACT-G (Functional Assessment of Cancer Therapy - General) Total Score From Baseline to 3 Months
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire that has four areas of measurements (physical well-being, social/family well-being, emotional well-being and functional well-being) with a scale of 0-4. The FACT-G total score ranges between 0 and 108. The higher the score, the better the quality of life. Change in FACT-G total score from baseline to 3 months was calculated as month 3 score - baseline score.
Time Frame: Assessed at baseline and 3 months
Population: Patients with baseline and 3-month FACT-G assessments were included in this analysis. Pediatric patients did not participate in the quality of life part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP)
Number analyzed (Participants) | 110 | 114 | 97
score on a scale | -4.9 (14.1) | -12.9 (14.1) | -3.4 (13.2)

6. Secondary Outcome: Change in FACIT-D (Functional Assessment of Cancer Therapy - Diarrhea) Diarrhea Subscale Score From Baseline to 3 Months
Description: The diarrhea subscale of The Functional Assessment of Chronic Illness Therapy - Diarrhea (FACIT-D) is an 11-item questionnaire with a scale of 0-4. The FACIT-D diarrhea subscale score ranges between 0 and 44. The higher the score, the better the quality of life. Change in FACIT-D diarrhea subscale score from baseline to 3 months was calculated as month 3 score - baseline score.
Time Frame: Assessed at baseline and 3 months
Population: Patients with baseline and 3-month FACIT-D diarrhea subscale assessments were included in this analysis. Pediatric patients did not participate in the quality of life part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP)
Number analyzed (Participants) | 109 | 114 | 97
score on a scale | -3.7 (6.9) | -0.7 (2.7) | -2.2 (5.1)

7. Secondary Outcome: Change in FACT-BRM (Functional Assessment of Cancer Therapy - Biologic Response Modifiers) Total Score From Baseline to 3 Months
Description: The Functional Assessment of Cancer Therapy - Biologic Response Modifiers (FACT-BRM) is a questionnaire including FACT-G (The Functional Assessment of Cancer Therapy - General) and additional sections addressing physical and mental quality of life aspects. It is a 40-item questionnaire with a scale of 0-4. The FACT-BRM total score ranges between 0 and 160. The higher the score, the better the quality of life. Change in FACT-BRM total score from baseline to 3 months is calculated as month 3 score - baseline score.
Time Frame: Assessed at baseline and 3 months
Population: Patients with baseline and 3-month FACT-BRM assessments were included in this analysis. Pediatric patients did not participate in the quality of life part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP)
Number analyzed (Participants) | 110 | 114 | 97
score on a scale | -8.3 (19.7) | -22.7 (20.4) | -6.2 (18.9)

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 20 years
Description: Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Groups:
- Arm D (HIP; Pediatric): Patients receive induction high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance high-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm E (HDI; Pediatric): Patients receive high-dose recombinant interferon alpha-2b IV on days 1-5, 8-12, 15-19, and 22-26 in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance high-dose recombinant interferon alpha-2b SC on days 1, 3, and 5. Treatment repeats every week for 48 weeks in the absence of disease progression or unacceptable toxicity.
- Arm F (LIP; Pediatric): Patients receive induction low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on week 24, patients receive maintenance low-dose ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (HIP) | Arm B (HDI) | Arm C (LIP) | Arm D (HIP; Pediatric) | Arm E (HDI; Pediatric) | Arm F (LIP; Pediatric)
All-Cause Mortality (participants affected / at risk) | 153/511 | 168/636 | 135/523 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 292/503 | 410/520 | 197/516 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 495/503 | 510/520 | 488/516 | 0/1 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (HIP) (N=503) | Arm B (HDI) (N=520) | Arm C (LIP) (N=516) | Arm D (HIP; Pediatric) (N=1) | Arm E (HDI; Pediatric) (N=1) | Arm F (LIP; Pediatric) (N=1)
Hearing impaired (Ear and labyrinth disorders) | 2 | 1 | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 5 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 26 | 120 | 14 | 0 | 0 | 0
Fever (General disorders) | 6 | 4 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 1 | 14 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0 | 11 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 40 | 5 | 23 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 18 | 0 | 12 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 5 | 1 | 3 | 0 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 43 | 0 | 20 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 4 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 52 | 1 | 35 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 6 | 0 | 5 | 0 | 0 | 0
Colonic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 73 | 4 | 54 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 0 | 6 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 19 | 25 | 5 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 5 | 2 | 1 | 0 | 0 | 0
Peritoneal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 13 | 12 | 3 | 0 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 16 | 2 | 5 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 5 | 0 | 2 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 3 | 0 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 5 | 2 | 2 | 0 | 0 | 0
Meningitis (Infections and infestations) | 4 | 0 | 2 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 1 | 3 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 40 | 78 | 15 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 4 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 32 | 61 | 11 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 6 | 2 | 2 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
CPK increased (Investigations) | 1 | 31 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 3 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 23 | 4 | 18 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 65 | 7 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 206 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 4 | 2 | 0 | 0 | 0
Serum amylase increased (Investigations) | 2 | 0 | 5 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 6 | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 70 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 3 | 0 | 3 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 13 | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 19 | 8 | 7 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 10 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 9 | 6 | 4 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 17 | 6 | 10 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 29 | 7 | 0 | 0 | 0
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 11 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 16 | 15 | 12 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 3 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 4 | 0 | 0 | 0
Syncope (Nervous system disorders) | 6 | 9 | 3 | 0 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 7 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 17 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psychosis (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 3 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 9 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 5 | 6 | 4 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (HIP) (N=503) | Arm B (HDI) (N=520) | Arm C (LIP) (N=516) | Arm D (HIP; Pediatric) (N=1) | Arm E (HDI; Pediatric) (N=1) | Arm F (LIP; Pediatric) (N=1)
Anemia (Blood and lymphatic system disorders) | 90 | 209 | 69 | NA | NA | NA
Chills (General disorders) | 61 | 178 | 34 | NA | NA | NA
Fatigue (General disorders) | 328 | 456 | 298 | NA | NA | NA
Fever (General disorders) | 98 | 174 | 53 | NA | NA | NA
Flu like symptoms (General disorders) | 39 | 254 | 34 | NA | NA | NA
Malaise (General disorders) | 10 | 31 | 6 | NA | NA | NA
Pain (General disorders) | 6 | 31 | 11 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 115 | 8 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 51 | 17 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 226 | 84 | 215 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 281 | 98 | 229 | NA | NA | NA
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 27 | 35 | 19 | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 61 | 3 | 42 | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 31 | 17 | 21 | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 103 | 50 | 54 | NA | NA | NA
Endocrine disorders - Other, specify (Endocrine disorders) | 94 | 12 | 65 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 103 | 39 | 89 | NA | NA | NA
Colitis (Gastrointestinal disorders) | 29 | 0 | 17 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 44 | 110 | 36 | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 234 | 176 | 231 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 20 | 88 | 14 | NA | NA | NA
Mucositis oral (Gastrointestinal disorders) | 16 | 35 | 7 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 182 | 361 | 147 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 83 | 133 | 54 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 140 | 342 | 86 | NA | NA | NA
Alkaline phosphatase increased (Investigations) | 53 | 42 | 26 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 125 | 367 | 72 | NA | NA | NA
Blood bilirubin increased (Investigations) | 24 | 48 | 22 | NA | NA | NA
CPK increased (Investigations) | 3 | 176 | 3 | NA | NA | NA
Lipase increased (Investigations) | 48 | 9 | 44 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 32 | 169 | 53 | NA | NA | NA
Neutrophil count decreased (Investigations) | 13 | 317 | 19 | NA | NA | NA
Platelet count decreased (Investigations) | 32 | 278 | 25 | NA | NA | NA
Serum amylase increased (Investigations) | 26 | 9 | 22 | NA | NA | NA
Weight loss (Investigations) | 57 | 214 | 35 | NA | NA | NA
White blood cell decreased (Investigations) | 12 | 273 | 15 | NA | NA | NA
Investigations - Other, specify (Investigations) | 107 | 95 | 91 | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 102 | 288 | 73 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 20 | 34 | 11 | NA | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 39 | 18 | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 | 51 | 31 | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 25 | 90 | 17 | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 32 | 52 | 21 | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 36 | 24 | 24 | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 17 | 93 | 18 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 | 102 | 44 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 27 | 8 | NA | NA | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 20 | 31 | 8 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 154 | 23 | NA | NA | NA
Dizziness (Nervous system disorders) | 45 | 109 | 25 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 21 | 165 | 16 | NA | NA | NA
Headache (Nervous system disorders) | 152 | 238 | 122 | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 43 | 25 | NA | NA | NA
Blurred vision (Eye disorders) | 37 | 29 | 15 | NA | NA | NA
Anxiety (Psychiatric disorders) | 15 | 93 | 14 | NA | NA | NA
Depression (Psychiatric disorders) | 20 | 160 | 17 | NA | NA | NA
Insomnia (Psychiatric disorders) | 28 | 92 | 25 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 42 | 17 | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 | 69 | 18 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT01274338/Prot_SAP_000.pdf